CLINICAL TRIAL: NCT06646328
Title: Oxidative Stress and Circulating Nuclear DNA (cfDNA) in Acute Kidney Injury and Continuous Renal Replacement Therapies. Effect of Two Anticoagulation Strategies of the Extracorporeal Purification System in Renal Function Recovery.
Brief Title: Oxidative Stress and Circulating Nuclear DNA (cfDNA) in Acute Kidney Injury and Continuous Renal Replacement Therapies.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment slower than anticipated and interrupted by COVID-19 pandemic
Sponsor: Fernando Sanchez (Other)
Collaborators: Hospital Universitario de la Plana (Other); Hospital General Universitario de Castellón (Other)
Responsible Party: Sponsor-Investigator, Fernando Sanchez, Consultant of Intensive Care Medicine, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FER-CIT-2016-01; 2016-004361-12 (EudraCT Number)
Record Dates: First submitted 2018-07-31; First posted 2024-10-17 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
Keywords: Biocompatibility; Renal replacement therapies; Oxidative stress; Myeloperoxidase; Nucleosomes; Regional citrate anticoagulation; Heparin
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy; Heparin; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparin (Active Comparator): Central venous access will be achieved with a 13 Fr double lumen catheter placed into the internal jugular or femoral vein.
  The patient will be connected to the Fresenius multiFiltrate (Fresenius Medical Care GmbH, Bad Homburg v.d.H., Germany) pump-assisted circuit with a high-flux synthetic membrane. In the heparin arm the anticoagulation technique to be used will be non-fractional heparin.
  Blood and ultrafiltrate samples will be taken from the prefilter (inlet filter plasma concentration [Ci]) and postfilter (outlet filter plasma concentration [Co]) sites of the extracorporeal circulation circuit at different times.
  Interventions: Procedure: Central venous access; Device: Pump-assisted circuit; Drug: Heparin sodium; Procedure: Blood and ultrafiltrate samples
- Citrate (Experimental): Central venous access will be achieved with a 13 Fr double lumen catheter placed into the internal jugular or femoral vein.
  The patient will be connected to the Fresenius multiFiltrate (Fresenius Medical Care GmbH, Bad Homburg v.d.H., Germany) pump-assisted circuit with a high-flux synthetic membrane. In the citrate arm regional citrate anticoagulation of the extracorporeal purification system will be used to avoid coagulation of the circuit.
  Blood and ultrafiltrate samples will be taken from the prefilter (inlet filter plasma concentration [Ci]) and postfilter (outlet filter plasma concentration [Co]) sites of the extracorporeal circulation circuit at different times.
  Interventions: Procedure: Central venous access; Device: Pump-assisted circuit; Other: Regional citrate anticoagulation; Procedure: Blood and ultrafiltrate samples

INTERVENTIONS:
Procedure: Central venous access — Venous access will be achieved with a 13 Fr double lumen catheter into the internal jugular or femoral vein.
Device: Pump-assisted circuit — The pump-assisted circuit to be used will be Fresenius multiFiltrate (Fresenius Medical Care GmbH, Bad Homburg v.d.H., Germany). EMIC2® Fresenius Medical Care high-flux synthetic membrane will be used
  Other Names: Continuous renal replacement therapy; CRRT
Drug: Heparin sodium — Non-fractional heparin will be used in one arm with an initial dose of 500-1000 IU/hour with adaptation of the infusion to the patient and the clotting time.
  Other Names: Non-fractional heparin; Heparin
  Arms: Heparin
Other: Regional citrate anticoagulation — Regional citrate anticoagulation will be used in the other arm with an initial dose of 3 mmol/L and with a calcium reinfusion solution at an initial dose of 2 mmol/L, with adaptation of both infusions to the patient ionic calcium levels.
  Arms: Citrate
Procedure: Blood and ultrafiltrate samples — Blood samples will be taken from the prefilter (inlet filter plasma concentration [Ci]) and postfilter (outlet filter plasma concentration [Co]) sites of the extracorporeal circulation circuit. The ultrafiltrate will be collected directly from the outlet of the hemofilter (ultrafiltrate concentration [Cuf]).
  The samples will taken at the beginning of CRRT (T0) and at the following times: T0, Ci; after 60 min (T1) and after 24 hours (T2) of CRRT, Ci, Co and Cuf.
  Venous access will be achieved with a 13 Fr double lumen catheter into the internal jugular or femoral vein.

SUMMARY:
Acute kidney injury (AKI) is the inability of the kidneys to perform their functions of purifying and cleaning the blood. It is a frequent complication in hospitalized patients, especially in those admitted to the ICUs. In these situations is common to use machines to artificially and temporarily replace renal function so waste products that can be toxic are removed from the body.

The purpose of this study is to assess the effectiveness and safety of two anticoagulation strategies of the extracorporeal purification system in critically ill patients with acute kidney injury treated with continuous renal replacement therapy (CRRT) evaluating the effect of both strategies in oxidative stress and extracellular nucleosomes and its influence on the recovery of renal function.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is defined as a sudden deterioration of renal function that causes loss of electrolyte control, acid base status and fluid balance, with subsequent accumulation of nitrogenous waste products that should be eliminated by the kidney. It is a frequent complication in hospitalized patients, especially those admitted to Intensive Care Units (ICUs). Its etiology is usually multifactorial, usually in the context of multiorgan dysfunction syndrome (MODS). The epidemiology and risk factors associated with its development, as well as the type of treatment that these patients are currently undergoing, continues to be the subject of debate, given the impact it has on morbidity and mortality.

To temporary substitute renal function in critically ill patients continuous renal replacement therapies (CRRT) are frequently used. The classification and nomenclature of techniques depends on the duration, continuity and operational characteristics of the treatment system. Thus, we distinguish between continuous techniques and intermittent techniques. Peritoneal dialysis (PD) is rarely used in developed countries for the treatment of AKI in ICU. Intermittent hemodialysis (IHD) is the most frequently used technique, although its use in ICU has considerable limitations on fluid balance, uremia control and elimination of medium molecular weight molecules.

Due to the enormous difficulty of obtaining studies with the necessary statistical power to provide the degree of evidence needed to clarify questions regarding the indications, modalities and other technical aspects of the CRRT, it is commonly used the experience that both the clinical practice in chronic patients as the results of scientific research that intermittent techniques (IHD fundamentally) confers to the clinician.

In patients with IHD, certain conditions are associated with a worse prognosis and an increased risk of mortality. These can include cardiovascular diseases, diabetes mellitus (DM), atherosclerosis, infectious processes, malnutrition, inflammation, oxidative stress, iron deficiency, anemia, calcification, uremia and volume overload. AKI requiring a renal replacement technique (RRT) represents an independent risk factor for mortality in critically ill patients. Oxidative stress and inflammation play important roles in the initiation and extension phases of AKI, as well as in causing injury to distant organs after AKI.

In CRRT to prevent coagulation of the extracorporeal system requires the use of some method of anticoagulation. The most frequent anticoagulation strategies include systemic heparin and regional citrate administration. However, some undesirable effects of CRRT may affect the patient's outcome, including the risks of systemic bleeding and membrane biocompatibility induced by anticoagulants.

Heparin, the most widely used anticoagulant in these techniques, is considered the standard of treatment, however it is contraindicated in patients with a high hemorrhagic risk or in heparin-induced thrombocytopenia.

Regional citrate anticoagulation (RCA), in which only the extracorporeal circuit is anticoagulated by the chelating action of calcium by citrate, is a safe and effective alternative in these cases. RCA has also been described as superior to heparin in terms of biocompatibility, since heparin, in comparison with citrate, can activate the complement and induce neutrophil degranulation in the filter and activate the release of myeloperoxidase (MPO) from the endothelium. The use of citrate, in addition to providing greater biocompatibility and a similar or longer filter duration, could also be associated with less inflammation and possibly with a better survival compared to heparin use, and probably also with a better renal recovery.

Apoptosis is probably implicated as a pathophysiological mechanism in organ injury in the setting of sepsis and systemic inflammatory response syndrome.

The sum effect of the numerous risk factors present in critical patients with AKI treated with CRRT is cumulative, additive, interrelated, complex and often unexpected or completely unknown. Survival in patients with AKI requiring replacement therapy is lower than in other patient populations. At present the accuracy of prediction of mortality and morbidity depending on available biomarkers or clinical condition is not optimal to properly describe and stratify patients properly. The combination of several markers of simultaneous biochemical processes can help to better stratify patients, identify the best therapeutic targets, evaluate the response to different therapies and establish functional prognoses. The usefulness of a parameter that evaluates tissue damage with markers of specific biochemical processes could be considered.

The present randomized, controlled, parallel-group, single centre study aims to evaluate the biocompatibility of two strategies of anticoagulation of the extracorporeal system (RCA and heparin) by using markers of inflammation, oxidative stress and cellular damage and its repercussion in the recovery of renal function. In this setting it would be possible to establish functional prognoses in terms of renal function recovery and to better identify which strategy is most beneficial for each group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients (age > 18) admitted to the ICU with AKI requiring treatment with continuous renal replacement technique.
* Patients able to accept being included in the study by signing the Informed Consent (IC). If the patient can not give consent, family consent is requested and, by default, the opinion of the person of trust or designated decision, if present. If there is no family present, trusted person or legal representative designated, the possibility of deferred consent is not contemplated. In this case the patient will not be included in the study.

Exclusion Criteria:

* Age under 18 years old.
* Pregnancy and/or lactation.
* Terminal diseases or life expectancy lower than 48 hours.
* Increased risk of bleeding (defined as platelet count less than 40x109 / L, partial thromboplastin time (TTPA) over 60 seconds, prothrombin time (PT)international normalized ratio (INR) greater than 2.0 or recent major bleeding).
* Need of systemic anticoagulation therapy.
* Contraindication for heparin.
* Heparin-induced Thrombocytopenia (HIT).
* Dialysis in the 24 hours prior to inclusion.
* Hypercalcemia (> 3 mmol / L).
* Severe Hepatitis: glutamic oxaloacetic transaminase (GOT) or glutamic pyruvic transaminase (GPT) > 1000 IU / L.
* Cirrhosis.
* Inclusion in another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Recovery of renal function | Through study completion, an average of 20 days.
  Impact of circulating nuclear DNA (cfDNA) and oxidative stress on duration of renal replacement therapy (RRT) in ICU.
Recovery of renal function | Through study completion, an average of 20 days.
  Impact of circulating nuclear DNA (cfDNA) and oxidative stress on change of Creatinine from baseline to ICU discharge.
Recovery of renal function | Through study completion, an average of 20 days.
  Impact of circulating nuclear DNA (cfDNA) and oxidative stress on change of Creatinine from baseline to hospital discharge.

SECONDARY OUTCOMES:
Activation and elimination of free radicals | 24 hours
  Changes in plasma concentration of glutathione (GSH) from baseline (before the initiation of the therapy) to 24 hours after de initiation of the therapy.
Activation and elimination of free radicals | 24 hours
  Changes in plasma concentration of glutathione disulfide (GSSG) from baseline (before the initiation of the therapy) to 24 hours after de initiation of the therapy.
Activation and elimination of biomarkers of inflammation | 24 hours
  Changes in plasma concentration of mieloperoxidase (MPO) from baseline (before the initiation of the therapy) to 24 hours after de initiation of the therapy.
Activation and elimination of biomarkers of inflammation | 24 hours
  Changes in plasma concentration of c-reactive protein (CRP) from baseline (before the initiation of the therapy) to 24 hours after de initiation of the therapy.
Activation and elimination of biomarkers of cell damage | 24 hours
  Changes in plasma concentration of circulating nuclear DNA (cfDNA) from baseline (before the initiation of the therapy) to 24 hours after de initiation of the therapy.
Mass transfer and clearance of free radicals | 24 hours
  Changes in plasma concentration of glutathione (GSH) from before to after the passage of blood through the filter
Mass transfer and clearance of free radicals | 24 hours
  Changes in plasma concentration of glutathione disulfide (GSSG) from before to after the passage of blood through the filter
Mass transfer and clearance of biomarkers of inflammation | 24 hours
  Changes in plasma concentration of mieloperoxidase (MPO) from before to after the passage of blood through the filter
Mass transfer and clearance of biomarkers of inflammation | 24 hours
  Changes in plasma concentration of c-reactive protein (CRP) from before to after the passage of blood through the filter
Mass transfer and clearance of biomarkers of cell damage | 24 hours
  Changes in plasma concentration of circulating nuclear DNA (cfDNA) from before to after the passage of blood through the filter
Length of stay | From ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 90 days
  Length of stay in ICU
Length of stay | From hospital admission until the date of documented hospital discharge or date of death from any cause, whichever came first, assessed up to 90 days
  Length of stay in hospital
Mortality | Through study completion, an average of 20 days.
  ICU mortality
Mortality | Day 90 after ICU admission
  Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Sanchez, MD, Study Chair — La Plana Health Department. Valencian Health Counseling; Fernando Sanchez, MD, Study Director — La Plana Health Department. Valencian Health Counseling; Fernando Sanchez, MD, Principal Investigator — La Plana Health Department. Valencian Health Counseling
Locations (1):
- Fernando Sánchez, Castellon, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hetzel GR, Schmitz M, Wissing H, Ries W, Schott G, Heering PJ, Isgro F, Kribben A, Himmele R, Grabensee B, Rump LC. Regional citrate versus systemic heparin for anticoagulation in critically ill patients on continuous venovenous haemofiltration: a prospective randomized multicentre trial. Nephrol Dial Transplant. 2011 Jan;26(1):232-9. doi: 10.1093/ndt/gfq575. Epub 2010 Sep 27. PMID 20876598
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Mehta RL, Chertow GM. Acute renal failure definitions and classification: time for change? J Am Soc Nephrol. 2003 Aug;14(8):2178-87. doi: 10.1097/01.asn.0000079042.13465.1a. No abstract available. PMID 12874474
- [Background] Herrera-Gutierrez ME, Seller-Perez G, Maynar-Moliner J, Sanchez-Izquierdo-Riera JA; Grupo de trabajo "Estado actual del fracaso renal agudo y de las tecnicas de reemplazo renal en UCI. Estudio FRAMI". [Epidemiology of acute kidney failure in Spanish ICU. Multicenter prospective study FRAMI]. Med Intensiva. 2006 Aug-Sep;30(6):260-7. doi: 10.1016/s0210-5691(06)74522-3. Spanish. PMID 16949000
- [Background] Liaño F, Candela A, Tenorio MT, Rodríguez-Palomares JR. La IRA en la UCI: Concepto, clasificaciones funcionales, epidemiología, biomarcadores, diagnóstico diferencial y pronóstico. En: Poch E, Liaño F, Gaínza F, eds. Manejo de la disfunción aguda del riñón del paciente crítico en la práctica clínica (primera ed.). Madrid: Ergon; 2011. pp. 1-21.
- [Background] Behrend T, Miller SB. Acute renal failure in the cardiac care unit: etiologies, outcomes, and prognostic factors. Kidney Int. 1999 Jul;56(1):238-43. doi: 10.1046/j.1523-1755.1999.00522.x. PMID 10411698
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Bellomo R, Ronco C, Mehta R. Nomenclature for continuous renal replacement therapies. Am J Kidney Dis. 1996;28(suppl 3):S2-S7.
- [Background] Liao Z, Zhang W, Hardy PA, Poh CK, Huang Z, Kraus MA, Clark WR, Gao D. Kinetic comparison of different acute dialysis therapies. Artif Organs. 2003 Sep;27(9):802-7. doi: 10.1046/j.1525-1594.2003.07282.x. PMID 12940902
- [Background] Alvestrand A, Ledebo I, Hagerman I, Wingren K, Mattsson E, Qureshi AR, Gutierrez A. Left ventricular hypertrophy in incident dialysis patients randomized to treatment with hemofiltration or hemodialysis: results from the ProFil study. Blood Purif. 2011;32(1):21-9. doi: 10.1159/000323140. Epub 2011 Jan 21. PMID 21252503
- [Background] Block GA, Hulbert-Shearon TE, Levin NW, Port FK. Association of serum phosphorus and calcium x phosphate product with mortality risk in chronic hemodialysis patients: a national study. Am J Kidney Dis. 1998 Apr;31(4):607-17. doi: 10.1053/ajkd.1998.v31.pm9531176.
- [Background] Degoulet P, Legrain M, Reach I, Aime F, Devries C, Rojas P, Jacobs C. Mortality risk factors in patients treated by chronic hemodialysis. Report of the Diaphane collaborative study. Nephron. 1982;31(2):103-10. doi: 10.1159/000182627. PMID 7121651
- [Background] Lonnemann G. Chronic inflammation in hemodialysis: the role of contaminated dialysate. Blood Purif. 2000;18(3):214-23. doi: 10.1159/000014420. PMID 10859424
- [Background] Panichi V, Rosati A, Bigazzi R, Paoletti S, Mantuano E, Beati S, Marchetti V, Bernabini G, Grazi G, Rizza GM, Migliori M, Giusti R, Lippi A, Casani A, Barsotti G, Tetta C; RISCAVID Study Group. Anaemia and resistance to erythropoiesis-stimulating agents as prognostic factors in haemodialysis patients: results from the RISCAVID study. Nephrol Dial Transplant. 2011 Aug;26(8):2641-8. doi: 10.1093/ndt/gfq802. Epub 2011 Feb 16. PMID 21325348
- [Background] Metnitz PG, Krenn CG, Steltzer H, Lang T, Ploder J, Lenz K, Le Gall JR, Druml W. Effect of acute renal failure requiring renal replacement therapy on outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2051-8. doi: 10.1097/00003246-200209000-00016. PMID 12352040
- [Background] Feltes CM, Van Eyk J, Rabb H. Distant-organ changes after acute kidney injury. Nephron Physiol. 2008;109(4):p80-4. doi: 10.1159/000142940. Epub 2008 Sep 18. PMID 18802379
- [Background] Tiranathanagul K, Jearnsujitwimol O, Susantitaphong P, Kijkriengkraikul N, Leelahavanichkul A, Srisawat N, Praditpornsilpa K, Eiam-Ong S. Regional citrate anticoagulation reduces polymorphonuclear cell degranulation in critically ill patients treated with continuous venovenous hemofiltration. Ther Apher Dial. 2011 Dec;15(6):556-64. doi: 10.1111/j.1744-9987.2011.00996.x. PMID 22107692
- [Background] Alonso A, Lau J, Jaber BL. Biocompatible hemodialysis membranes for acute renal failure. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD005283. doi: 10.1002/14651858.CD005283. PMID 15846749
- [Background] Oudemans-van Straaten HM, Kellum JA, Bellomo R. Clinical review: anticoagulation for continuous renal replacement therapy--heparin or citrate? Crit Care. 2011 Jan 24;15(1):202. doi: 10.1186/cc9358. PMID 21345279
- [Background] Palsson R, Niles JL. Regional citrate anticoagulation in continuous venovenous hemofiltration in critically ill patients with a high risk of bleeding. Kidney Int. 1999 May;55(5):1991-7. doi: 10.1046/j.1523-1755.1999.00444.x. PMID 10231464
- [Background] Nurmohamed SA, Vervloet MG, Girbes AR, Ter Wee PM, Groeneveld AB. Continuous venovenous hemofiltration with or without predilution regional citrate anticoagulation: a prospective study. Blood Purif. 2007;25(4):316-23. doi: 10.1159/000107045. Epub 2007 Aug 14. PMID 17700015
- [Background] Schilder L, Nurmohamed SA, ter Wee PM, Paauw NJ, Girbes AR, Beishuizen A, Beelen RH, Groeneveld AB. Citrate confers less filter-induced complement activation and neutrophil degranulation than heparin when used for anticoagulation during continuous venovenous haemofiltration in critically ill patients. BMC Nephrol. 2014 Jan 17;15:19. doi: 10.1186/1471-2369-15-19. PMID 24438360
- [Background] Oudemans-van Straaten HM, Bosman RJ, Koopmans M, van der Voort PH, Wester JP, van der Spoel JI, Dijksman LM, Zandstra DF. Citrate anticoagulation for continuous venovenous hemofiltration. Crit Care Med. 2009 Feb;37(2):545-52. doi: 10.1097/CCM.0b013e3181953c5e. PMID 19114912
- [Background] Schneider AG, Bagshaw SM. Effects of renal replacement therapy on renal recovery after acute kidney injury. Nephron Clin Pract. 2014;127(1-4):35-41. doi: 10.1159/000363671. Epub 2014 Sep 24. PMID 25343818
- [Background] Zhang Z, Hongying N. Efficacy and safety of regional citrate anticoagulation in critically ill patients undergoing continuous renal replacement therapy. Intensive Care Med. 2012 Jan;38(1):20-8. doi: 10.1007/s00134-011-2438-3. Epub 2011 Nov 29. PMID 22124775
- [Background] Kellum JA, Bellomo R, Mehta R, Ronco C. Blood purification in non-renal critical illness. Blood Purif. 2003;21(1):6-13. doi: 10.1159/000067862. PMID 12566655
- [Background] Rimmele T, Kellum JA. Clinical review: blood purification for sepsis. Crit Care. 2011;15(1):205. doi: 10.1186/cc9411. Epub 2011 Feb 16. PMID 21371356
- [Background] Hotchkiss RS, Swanson PE, Freeman BD, Tinsley KW, Cobb JP, Matuschak GM, Buchman TG, Karl IE. Apoptotic cell death in patients with sepsis, shock, and multiple organ dysfunction. Crit Care Med. 1999 Jul;27(7):1230-51. doi: 10.1097/00003246-199907000-00002. PMID 10446814
- [Background] Lerolle N, Nochy D, Guerot E, Bruneval P, Fagon JY, Diehl JL, Hill G. Histopathology of septic shock induced acute kidney injury: apoptosis and leukocytic infiltration. Intensive Care Med. 2010 Mar;36(3):471-8. doi: 10.1007/s00134-009-1723-x. PMID 19924395
- [Background] Niu G, Chen X. Apoptosis imaging: beyond annexin V. J Nucl Med. 2010 Nov;51(11):1659-62. doi: 10.2967/jnumed.110.078584. Epub 2010 Oct 18. PMID 20956479
- [Background] Atan R, Virzi GM, Peck L, Ramadas A, Brocca A, Eastwood G, Sood S, Ronco C, Bellomo R, Goehl H, Storr M. High cut-off hemofiltration versus standard hemofiltration: a pilot assessment of effects on indices of apoptosis. Blood Purif. 2014;37(4):296-303. doi: 10.1159/000363220. Epub 2014 Aug 1. PMID 25096908
- [Background] Bortner CD, Oldenburg NB, Cidlowski JA. The role of DNA fragmentation in apoptosis. Trends Cell Biol. 1995 Jan;5(1):21-6. doi: 10.1016/s0962-8924(00)88932-1. PMID 14731429
- [Background] Zeerleder S, Zwart B, Wuillemin WA, Aarden LA, Groeneveld AB, Caliezi C, van Nieuwenhuijze AE, van Mierlo GJ, Eerenberg AJ, Lammle B, Hack CE. Elevated nucleosome levels in systemic inflammation and sepsis. Crit Care Med. 2003 Jul;31(7):1947-51. doi: 10.1097/01.CCM.0000074719.40109.95. PMID 12847387
- [Background] Chen Q, Ye L, Jin Y, Zhang N, Lou T, Qiu Z, Jin Y, Cheng B, Fang X. Circulating nucleosomes as a predictor of sepsis and organ dysfunction in critically ill patients. Int J Infect Dis. 2012 Jul;16(7):e558-64. doi: 10.1016/j.ijid.2012.03.007. Epub 2012 May 18. PMID 22609014
- [Background] Butt AN, Swaminathan R. Overview of circulating nucleic acids in plasma/serum. Ann N Y Acad Sci. 2008 Aug;1137:236-42. doi: 10.1196/annals.1448.002. PMID 18837954
- [Background] Garcia Moreira V, de la Cera Martinez T, Gago Gonzalez E, Prieto Garcia B, Alvarez Menendez FV. Increase in and clearance of cell-free plasma DNA in hemodialysis quantified by real-time PCR. Clin Chem Lab Med. 2006;44(12):1410-5. doi: 10.1515/CCLM.2006.252. PMID 17163815
- [Background] Tovbin D, Novack V, Wiessman MP, Abd Elkadir A, Zlotnik M, Douvdevani A. Circulating cell-free DNA in hemodialysis patients predicts mortality. Nephrol Dial Transplant. 2012 Oct;27(10):3929-35. doi: 10.1093/ndt/gfs255. Epub 2012 Jul 24. PMID 22833622
- [Background] Boschetti-de-Fierro A, Voigt M, Storr M, Krause B. Extended characterization of a new class of membranes for blood purification: the high cut-off membranes. Int J Artif Organs. 2013 Jul;36(7):455-63. doi: 10.5301/ijao.5000220. Epub 2013 May 10. PMID 23661558
- [Background] Atan R, Crosbie DC, Bellomo R. Techniques of extracorporeal cytokine removal: a systematic review of human studies. Ren Fail. 2013 Sep;35(8):1061-70. doi: 10.3109/0886022X.2013.815089. Epub 2013 Jul 19. PMID 23866032
- [Background] Atan R, May C, Bailey SR, Tanudji M, Visvanathan K, Skinner N, Bellomo R, Goehl H, Storr M. Nucleosome levels and toll-like receptor expression during high cut-off haemofiltration: a pilot assessment. Crit Care Resusc. 2015 Dec;17(4):239-43. PMID 26640058
- [Background] Zeerleder S, Stephan F, Emonts M, de Kleijn ED, Esmon CT, Varadi K, Hack CE, Hazelzet JA. Circulating nucleosomes and severity of illness in children suffering from meningococcal sepsis treated with protein C. Crit Care Med. 2012 Dec;40(12):3224-9. doi: 10.1097/CCM.0b013e318265695f. PMID 22932399
- [Background] Kofoed K, Andersen O, Kronborg G, Tvede M, Petersen J, Eugen-Olsen J, Larsen K. Use of plasma C-reactive protein, procalcitonin, neutrophils, macrophage migration inhibitory factor, soluble urokinase-type plasminogen activator receptor, and soluble triggering receptor expressed on myeloid cells-1 in combination to diagnose infections: a prospective study. Crit Care. 2007;11(2):R38. doi: 10.1186/cc5723. PMID 17362525
- [Background] Punyadeera C, Schneider EM, Schaffer D, Hsu HY, Joos TO, Kriebel F, Weiss M, Verhaegh WF. A biomarker panel to discriminate between systemic inflammatory response syndrome and sepsis and sepsis severity. J Emerg Trauma Shock. 2010 Jan;3(1):26-35. doi: 10.4103/0974-2700.58666. PMID 20165718
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] KDIGO AKI Work Group. KDIGO clinical practice guideline for acute kidney injury. Kidney Int Suppl. 2012;17:1-138.
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Villa G, Neri M, Bellomo R, Cerda J, De Gaudio AR, De Rosa S, Garzotto F, Honore PM, Kellum J, Lorenzin A, Payen D, Ricci Z, Samoni S, Vincent JL, Wendon J, Zaccaria M, Ronco C; Nomenclature Standardization Initiative (NSI) Alliance. Nomenclature for renal replacement therapy and blood purification techniques in critically ill patients: practical applications. Crit Care. 2016 Oct 10;20(1):283. doi: 10.1186/s13054-016-1456-5. PMID 27719676
- [Background] Maynar-Moliner J, Sanchez-Izquierdo-Riera JA, Herrera-Gutierrez M. Renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Oct 30;359(18):1960; author reply 1961-2. No abstract available. PMID 18979570
- [Background] Maynar Moliner J, Honore PM, Sanchez-Izquierdo Riera JA, Herrera Gutierrez M, Spapen HD. Handling continuous renal replacement therapy-related adverse effects in intensive care unit patients: the dialytrauma concept. Blood Purif. 2012;34(2):177-85. doi: 10.1159/000342064. Epub 2012 Oct 24. PMID 23095418
- [Background] Honore PM, Jacobs R, Joannes-Boyau O, De Waele E, Van Gorp V, Boer W, Spapen HD. Con: Dialy- and continuous renal replacement (CRRT) trauma during renal replacement therapy: still under-recognized but on the way to better diagnostic understanding and prevention. Nephrol Dial Transplant. 2013 Nov;28(11):2723-7; discussion 2727-8. doi: 10.1093/ndt/gft086. PMID 24169609
- [Background] Link A, Klingele M, Speer T, Rbah R, Poss J, Lerner-Graber A, Fliser D, Bohm M. Total-to-ionized calcium ratio predicts mortality in continuous renal replacement therapy with citrate anticoagulation in critically ill patients. Crit Care. 2012 May 29;16(3):R97. doi: 10.1186/cc11363. PMID 22643456
- [Background] Slowinski T, Morgera S, Joannidis M, Henneberg T, Stocker R, Helset E, Andersson K, Wehner M, Kozik-Jaromin J, Brett S, Hasslacher J, Stover JF, Peters H, Neumayer HH, Kindgen-Milles D. Safety and efficacy of regional citrate anticoagulation in continuous venovenous hemodialysis in the presence of liver failure: the Liver Citrate Anticoagulation Threshold (L-CAT) observational study. Crit Care. 2015 Sep 29;19:349. doi: 10.1186/s13054-015-1066-7. PMID 26415638
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Liano F, Gallego A, Pascual J, Garcia-Martin F, Teruel JL, Marcen R, Orofino L, Orte L, Rivera M, Gallego N, et al. Prognosis of acute tubular necrosis: an extended prospectively contrasted study. Nephron. 1993;63(1):21-31. doi: 10.1159/000187139. PMID 8446248
- [Background] Oh H, Siano B, Diamond S. Neutrophil isolation protocol. J Vis Exp. 2008 Jul 23;(17):745. doi: 10.3791/745. PMID 19066523
- [Background] Chen G, Zhang D, Fuchs TA, Manwani D, Wagner DD, Frenette PS. Heme-induced neutrophil extracellular traps contribute to the pathogenesis of sickle cell disease. Blood. 2014 Jun 12;123(24):3818-27. doi: 10.1182/blood-2013-10-529982. Epub 2014 Mar 11. PMID 24620350
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- See also: SPAIN. 2015. BOE-A-2015-14082. Royal Decree 1090/2015, of December 4, regulating clinical trials with medicines, Committees of Ethics of Research with medicines and the Spanish Registry of Clinical Studies. — http://www.boe.es/boe/dias/2015/12/24/pdfs/BOE-A-2015-14082.pdf
- See also: EUROPEAN UNION. OJ L 158 27.5.2014. Regulation (EU) No 536/2014 of the European Parliament and of the Council of 16 April 2014 on clinical trials on medicinal products for human use and repealing Directive 2001/20 / EC. — http://data.europa.eu/eli/reg/2014/536/oj
- See also: SPAIN. 2007. BOE-A-2007-12945. Law 14/2007, of July 3, on Biomedical Research which regulates biomedical research. Official Gazette of the State, July 4, 2007, 159, pp. 28826 to 28848. — http://www.boe.es/boe/dias/2007/07/04/pdfs/A28826-28848.pdf